CLINICAL TRIAL: NCT01275053
Title: In Vivo Leptin Signaling in Humans After Acute Leptin Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Professor in Public Health, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002P000097
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Lean; Obese; Obese Diabetics
Keywords: Leptin; In Vivo; Diabetic; Obese; Lean
MeSH Terms: conditions — Obesity | interventions — Leptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Leptin (Experimental)
  Interventions: Drug: leptin

INTERVENTIONS:
Drug: leptin — 0.01mg/kg

SUMMARY:
The purpose of this research study is to help us to better understand how leptin regulates blood sugar levels. Leptin is a recently discovered hormone, which is made in fat cells. Leptin is secreted by fat and acts as a signal to the brain to decrease appetite and influences how the body regulates blood sugar levels. A synthetic form of leptin (A-100), an investigational drug and has not yet been approved by the Food and Drug Administration (FDA), will be administered to participants in this study. The expected duration of your participation is 3 study visits, which will be spread over 3-4 weeks.

This study involves having fat and muscle biopsies after receiving leptin under local anesthesia in the General Clinical Research Center (GCRC), surgical unit, and/or Endocrinology exam room at the Beth Israel Deaconess Medical Center.

DETAILED DESCRIPTION:
Screening Visit During this visit, you will have a complete medical history taken and have a physical examination performed by one of the study physicians. You will also have your height and weight measured. You will have a blood drawn (approximately 2 tablespoons)and will have an electrocardiogram (EKG). At the screening visit you will also meet with a dietician who will review your food preferences with you in order to design the meals that you will receive as part of the study.

Study Day #1: You will pick up your meals designed with the dietician. You will be provided with meals for 48 hours prior to your fat biopsy. These meals will be designed by the dietician based upon what you like to eat. You will also have your Resting Metabolic Rate Measured.

Study Day #2: A nurse will will insert two intravenous catheters (IV) into a medium size vein in each of your forearms. You will then have two fat and muscle thigh biopsy. One before and one after leptin is given. You will stay in the hospital for three hours of observation. During this time you will have your Resting Metabolic Rate measured and then you will be provided with a meal.

Study Day #3: Seven to ten days after the biopsy, you will be asked to return to the hospital so that the surgeon can inspect the wound.

Your participation in this study will involve 3 study visits, which will be spread out over 3-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* For this pilot study we propose to enroll men and women, ages 18-65 years, with body mass index (BMI) ranges meeting lean and obese criteria, and less than or equal to 45 kg/m2. Obese diabetics will also be included.

Exclusion Criteria:

* We will exclude subjects who require special diet prior to biopsy. We will exclude subjects with a history of any illness, other than obesity and diabetes. Subjects taking any medications that are known to influence glucose metabolism such as glucocorticoids will also be excluded. Subjects who have a known history of anaphylaxis or anaphylactoid-like reactions or who have a known hypersensitivity to E. coli-derived proteins or anesthetic agents such as Lidocaine or Novocaine will be excluded from the study. Women who are breast feeding, pregnant, or wanting to become pregnant during the month following the study may not participate in this study. Women participating in this study must use a contraceptive method to prevent pregnancy (birth control pills, hormonal implants, intrauterine device (IUD), diaphragm with intravaginal spermicide, cervical cap, male or female condom). If a woman suspects that she has become pregnant during the study or within one month of completing study, or if she does not use one of the contraceptive methods recommended by the investigator, she will be instructed to notify the study staff immediately. Subjects with a history of bleeding dyscrasia, poor wound healing or any medical condition precluding supine position will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2002-07; Primary Completion 2013-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos s Mantzoros, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matarese G, La Rocca C, Moon HS, Huh JY, Brinkoetter MT, Chou S, Perna F, Greco D, Kilim HP, Gao C, Arampatzi K, Wang Z, Mantzoros CS. Selective capacity of metreleptin administration to reconstitute CD4+ T-cell number in females with acquired hypoleptinemia. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):E818-27. doi: 10.1073/pnas.1214554110. Epub 2013 Feb 4. PMID 23382191

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leptin
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Leptin
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  All participants | 43.3 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Leptin Signaling
Description: Leptin signaling is assessed before and 30 minutes after in vivo metreleptin administration.
  The primary outcome was p-STAT3/STAT3 in biopsies (fat tissue) before and 30 minutes after in vivo metreleptin administration.
  The p-STAT3/STAT3 before metreleptin administration was given the value 1, and the p-STAT3/STAT3 30 minutes after in vivo metreleptin administration was given the value showing the fold change compared to p-STAT3/STAT3 before metreleptin administration.
Time Frame: Baseline and 30 minutes
Population: All subjects received biopsies before and 30 min after leptin administration.
Measure: Mean (Full Range); unit: fold change
Arm/Group | Leptin
Number analyzed (Participants) | 12
fold change | 3.1 [2.8 to 3.4]

ADVERSE EVENTS:
Arm/Group | Leptin
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No